CLINICAL TRIAL: NCT05297526
Title: Happy Teeth for Hopi Tots: Cultural Adaptation of an Oral Health Entertainment-Education Intervention to Prevent Early Childhood Caries Among American Indian Children
Brief Title: Happy Teeth for Hopi Tots: Cultural Adaptation of an Oral Health Entertainment-Education Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruite participants due to COVID-19 and other barriers
Sponsor: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Heather Thomas, Associate Clinical Professor, Northern Arizona University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1774258-2
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Early Childhood Caries
Keywords: Oral Health; Health Knowledge, Attitudes, Practice; Health Education, Dental; American Indian; Dental Caries; Cultural Adaptation
MeSH Terms: conditions — Behavior; Health Education; Dental Caries

STUDY DESIGN:
Intervention Model Description: After completing the consent and baseline survey, participants will be randomized into either the control group or the intervention group via Jefferson REDCap. Participants will not know which group they are in, and will receive the corresponding materials for their group to use for the duration of the study (3 months). At the end of the 3 month period, participants will take a post-study survey to gauge changes in knowledge, attitudes, and behaviors regarding oral health. At the end of the trial, participants who were in the control group receiving just the informational pamphlet, will receive a copy of the baby book given to the intervention group.
Who Masked: Participant
Masking Description: Participants will be masked as to which group they have been randomized into for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a culturally adapted children's book that contains the same oral health educational information as the control brochure, but celebrates Tribe-specific culture and utilizes entertainment education. The children's book includes vibrant illustrations by a Tribal artist, and has eBook and audio narration options for multi-media use and/or those with limited literacy.
  Interventions: Behavioral: Culturally adapted children's book
- Control Group (Active Comparator): The control group will receive a standard educational brochure about children's oral health designed by the the National Institutes for Health (NIH) for American Indian/Alaska Native parents.
  Interventions: Behavioral: Standard informational brochure on children's oral health

INTERVENTIONS:
Behavioral: Culturally adapted children's book — Tribe-specific children's book celebrating tribal culture with an embedded oral health message
  Other Names: Education entertainment
  Arms: Intervention Group
Behavioral: Standard informational brochure on children's oral health — Informational brochure about children's oral health designed by the NIH for American Indian/Alaska Native parents.
  Arms: Control Group

SUMMARY:
Tooth decay is a preventable disease occurring at high rates among American Indian (AI) populations. The use of entertaining educational materials and cultural adaptation have shown success in improving health behaviors. This trial will test changes in AI parents' knowledge, attitudes and behaviors related to their child(ren)'s oral health after utilizing a culturally adapted children's book/eBook, versus a standard oral health pamphlet developed by the NIH. I hypothesize that the parents in the intervention (book) group will exhibit greater improvement of these measures.

DETAILED DESCRIPTION:
Early childhood caries (ECC), or the presence of one or more decayed, missing, or filled teeth in children age 5 or younger, is the most chronic childhood disease though it is largely preventable. ECC is most prevalent among American Indian and Alaskan Native (AI/AN) children, with nearly 60% experiencing decay by the age of 3 and over 75% by the age of 5. Oral health is a significant indicator of overall well-being, health, and quality of life, and can have grave impacts on children and their families when disease is not addressed.

Dental decay in primary (baby) teeth can cause pain, damage to the permanent teeth, infection of the head and neck, and difficulty chewing. Severe decay can interfere with intellectual and social development, cause poor speech articulation, embarrassment, low self-esteem, missed days at school, and social isolation. In addition to the physical, psychosocial, and developmental toll on children and their families, treatment for ECC is costly, particularly when hospitalization and general anesthesia are required, which is often the case with severe decay. Because ECC is preventable and can progress quickly, early intervention is a key strategy in reducing its prevalence, particularly in high risk populations.

Interventions utilizing a variety of approaches to address ECC among AI/AN populations have produced mixed results, but few have explored the effect of creative cultural adaptation of oral health education materials on parental knowledge, attitudes, and behaviors regarding the oral health of their children. The use of Entertainment Education (E-E) and specific cultural adaptation of intervention materials have shown success in improving health behaviors of minority and disadvantaged populations. This project will utilize an experimental design using a convenience sample of Hopi parents/caregivers living off Tribal lands, who will be randomized into either the intervention group receiving a culturally adapted children's book celebrating tribal culture with an embedded oral health message, or the control group receiving a standard educational brochure developed by the National Institutes for Health (NIH) for AI/AN. The children's book has electronic book (eBook) and audio narration options for multi-media use and/or those with limited literacy and was illustrated and narrated by Tribal members. Formative assessment data from an ongoing NIH clinical trial involving AI mothers/caregivers and their children in the prevention of ECC (NCT04556175), including Hopi Tribal Community Advisory Board (CAB) meetings, and a review of current literature informed the development of intervention materials (children's book) for this study. The aim of this study is to test the impact of a culturally adapted oral health E-E intervention on the knowledge, attitudes and behaviors of American Indian parents/caregivers related to their child(ren)'s oral health.

The purpose of this research is to identify effective interdisciplinary avenues to reduce the incidence of ECC among AI/AN children. The objective of this study is to compare the effect of a culturally adapted Entertainment-Education intervention on AI parents' knowledge, attitudes, and behaviors pertaining to their children's oral health, to a standard educational brochure developed by the NIH for AI/AN parents.

The main outcome variables will be mean changes from baseline to follow-up in oral health knowledge, beliefs, and behaviors in the intervention group compared to the control group. Post-hoc analyses will be utilized to determine which specific outcome variables (i.e., knowledge, beliefs, or behavior) differed between the groups (primary outcomes).

I hypothesize the that the parents/caregivers in the intervention group will exhibit greater improvement of oral health knowledge, attitudes, and behavior than parents/caregivers in the control group who receive a standard informational pamphlet.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Be willing and able to follow study procedures and instructions for the duration of the study (3 months)
* Be at least 18 years of age
* Have access to the internet to complete the consent form, surveys and receive incentives for participation
* Provide a valid mailing address and email address to receive study materials and receive incentives
* Be a parent or caregiver of a child or children under the age of 6 years old.
* Be a member of the Hopi Tribe who does not live on Tribal lands. American Indian status is self-identified-no tribal enrollment verification will be required.
* Not be an enrolled member of the Navajo Tribe, AND
* Not be living on Hopi or Navajo Nations.

Exclusion Criteria:

* Are not able to understand or sign a consent form for yourself to participate
* Under 18 years of age
* Do not have access to the internet to complete surveys
* Do not provide a valid mailing address and email address to receive study materials and incentives
* Not a member of the Hopi Tribe
* An enrolled member of the Navajo Tribe
* Living on the Hopi or Navajo Nations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Oral Health Knowledge after 3 months Intervention | Three months from completion of baseline survey, each participant will fill out the post-study survey.
  Quantitative changes in knowledge attitudes, and behaviors will be measured using an adapted version of the Basic Research Factors Questionnaire (BRFQ), an instrument developed to assess common risk factors for ECC among high-risk populations (Albino, et al., 2017). The questionnaire will be administered before and after the 3-month intervention via the secure Jefferson REDCap online platform. Increases in oral health knowledge, positive attitudes and reported oral health behaviors indicate a positive outcome.
  Measures for Oral health knowledge of parents /caregivers [Time Frame: assessed at baseline and after 3 months.]
  Percentage of correct responses to 22 knowledge questions based on the BRFQ (Albino, et al., 2017). There are 11 true/false questions, 8 Likert-type judgements of whether certain behaviors are good for a child's teeth, and 3 multiple choice questions regarding infant/child oral health care. A higher percentage of correct responses indicates a better outcome.
Changes from Baseline in Oral Health Attitudes after 3 months Intervention | Three months from completion of baseline survey, each participant will fill out the post-study survey.
  Measures for Attitudes towards oral health care of parents /caregivers [ Time Frame: assessed at baseline and after 3 months.]
  Sum of Likert-type ratings (on a scale of 1-5) for 36 items regarding attitudes toward oral health care. Twenty-four of the items are based upon the Basic Research Factors Questionnaire (Albino, et al., 2017); 12 items measure the importance of oral health care and 12 measure parental/caregiver dental self-efficacy to adhere to oral health care. Twelve study-specific items were added to measure parental caregiver intention to perform the 12 items measured for importance and self-efficacy. Scores range from 36 (lowest) to 180 (highest) with higher scores representing more favorable attitudes towards child oral health care.
Changes from Baseline in Oral Health Behaviors after 3 months Intervention | Three months from completion of baseline survey, each participant will fill out the post-study survey.
  Measures for Oral health behavior of parents/caregivers [Time Frame: assessed at baseline and after 3 months.]
  Percentage of correct responses to 22 questions regarding oral health behavior based upon the Basic Research Factors Questionnaire (Albino, et al., 2017). Items include 8 questions regarding dental health care utilization, 10 questions regarding parental oral health care habits for self and child, and 4 questions regarding child's consumption of sweets/sugar. A higher percentage of correct responses indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Thomas, MEd, Principal Investigator — Northern Arizona University
Locations (1):
- Dental Hygiene Department, Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albino J, Tiwari T, Gansky SA, Henshaw MM, Barker JC, Brega AG, Gregorich SE, Heaton B, Batliner TS, Borrelli B, Geltman P, Kressin NR, Weintraub JA, Finlayson TL, Garcia RI; Early Childhood Caries Collaborating Centers. The basic research factors questionnaire for studying early childhood caries. BMC Oral Health. 2017 May 19;17(1):83. doi: 10.1186/s12903-017-0374-5. PMID 28526003